CLINICAL TRIAL: NCT05818176
Title: To Improve the Clinical Outcome of Ultrasound-guided Radiofrequency Ablation by NAVIRFA® Navigation System.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202211106DIPB
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Radiofrequency Ablation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAVIRFA® Navigation System (Experimental)
  Interventions: Device: NAVIRFA® Navigation System
- ultrasound-guided (Active Comparator)
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: NAVIRFA® Navigation System — radiofrequency ablation by NAVIRFA® Navigation System.
  Arms: NAVIRFA® Navigation System
Device: ultrasound — radiofrequency ablation by ultrasound
  Arms: ultrasound-guided

SUMMARY:
Ultrasonic-guided radiofrequency ablation is the most common minimally invasive treatment for liver cancer. This study will use my country's self-developed intelligent ultrasonic navigation tool (NAVIRFA® Navigation System) to assist in the puncture of the needle during ablation, to observe the operation time, Whether the needle accuracy, ablation effect and complications are different from the traditional free-hand ultrasonic guidance technology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malignant liver tumors less than three centimeters in size who are expected to suffer radiofrequency tumor ablation in the hospital.
2. At least 20 years old.

Exclusion Criteria:

1. Patients with abnormal coagulation function and low platelets are not suitable for ablation therapy after evaluation by the trial host.
2. Those who are unable to accept computerized tomography and MRI examinations, such as poor renal function or contrast agent allergy, are not suitable for examination after the evaluation of the test host.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
required scan time | Before ablation treatment
  the time required until start of the ablation (measured from the time of the first US scan to the start of the ablation).

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan